CLINICAL TRIAL: NCT00544765
Title: A Multi-center Randomized Phase III Study Evaluating 4 Cycles of Docetaxel, Doxorubicin and Cyclophosphamide Versus 4 Cycles of Vinorelbine and Capecitabine in Patients Not Sufficiently Responding to 2 Cycles of TAC and 4 Cycles of TAC Versus 6 Cycles of TAC in Patients Sufficiently Responding to 2 Cycles of TAC as Preoperative Treatment of Locally Advanced or Operable Primary Breast Cancer
Brief Title: Docetaxel, Doxorubicin and Cyclophosphamide Versus Vinorelbine and Capecitabine in Patients Not Sufficiently / Sufficiently Responding as Preoperative Treatment of Locally Advanced or Operable Primary Breast Cancer
Acronym: GeparTrio
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Roche Pharma AG (Industry); Sanofi (Industry); Amgen (Industry); Goethe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 24
Record Dates: First submitted 2007-07-20; First posted 2007-10-16 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; neoadjuvant therapy; pCR rates
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- resp: 4xTAC (Experimental): Patients sufficiently responding (iPR, iCR) will recieve 4 further cycles of TAC
  Interventions: Drug: TAC
- resp: 6xTAC (Experimental): Patients sufficiently responding (iPR, iCR) will recieve 6 further cycles of TAC
  Interventions: Drug: TAC
- nonResp: 4xTAC (Experimental): Patients non-sufficiently responding (iNC) will recieve 4 further cycles of TAC
  Interventions: Drug: TAC
- nonResp: 4xNX (Experimental): Patients non-sufficiently responding (iNC) will recieve 4 further cycles of NX
  Interventions: Drug: NX

INTERVENTIONS:
Drug: TAC — Docetaxel 75 mg/m² as a 1 hour i.v. infusion on day 1 every 3 weeks in combination with Doxorubicin 50 mg/m² as an i.v. bolus and Cyclophosphamide 500 mg/m2 as an i.v. bolus on day 1 every 3 weeks
  Arms: nonResp: 4xTAC; resp: 4xTAC; resp: 6xTAC
Drug: NX — Vinorelbine 25 mg/m² as a < 10 min i.v. infusion on days 1 and 8 repeated every 3 weeks and Capecitabine 2000 mg/m² orally in 2 daily doses on days 1-14 repeated every 3 weeks
  Arms: nonResp: 4xNX

SUMMARY:
Primary objective of the study in patients without a sufficient sonographic response (i.e. iNC) to 2 cycles of TAC as preoperative treatment of operable (T>/= 2cm, N0-2,M0) primary breast cancer: To determine the response rate determined by sonography (iRR = iCR+iPR) of further 4 cycles of docetaxel, doxorubicin and cyclophosphamide (TAC) and of 4 cycles of vinorelbine and capecitabine (NX) (TAC vs. NX)

Primary objective of the study in patients with a sufficient sonographic response (i.e. iRR = iPR or iCR) to the first 2 cycles of TAC as preoperative treatment of operable (T>/=2cm, N0-2,M0) primary breast cancer: To determine the pCR rate of 6 cycles vs. 8 cycles of docetaxel, doxorubicin and cyclophosphamide (TAC x 6 vs. TAC x 8)

DETAILED DESCRIPTION:
Prospective, randomized phase III trial Study population I: operable (T>/=2cm, N0-2,M0) primary breast cancer Study population II: locally advanced (T4 a-d, N0-3,M0) primary breast cancer patients

All patients will receive 2 cycles of TAC. Thereafter

* Patients sufficiently responding (iPR, iCR) will be randomized to either 4 further cycles of TAC or 6 further cycles of TAC
* Patients non-sufficiently responding (iNC) will be randomized to either 4 further cycles of TAC or 4 cycles of NX:

TAC: Docetaxel 75 mg/m² as a 1 hour i.v. infusion on day 1 every 3 weeks in combination with Doxorubicin 50 mg/m² as an i.v. bolus and Cyclophosphamide 500 mg/m2 as an i.v. bolus on day 1 every 3 weeks

NX: Vinorelbine 25 mg/m² as a 10 min i.v. infusion on days 1 and 8 repeated every 3 weeks and Capecitabine 2000 mg/m² orally in 2 daily doses on days 1-14 repeated every 3 weeks If a patient shows progressive disease during the first 2 cycles of TAC she will not be randomized and will be treated according to the discretion of the investigator. In patients with disease progression during further preoperative therapy, the treatment should be discontinued and patients should be treated by immediate surgery. In case of inoperability even after termination of chemotherapy further treatment is to the discretion of the investigator (e.g. radiotherapy).

Dose reduction and/or treatment delay and treatment discontinuation are planned in case of severe hematological and/or non-hematological toxicities.

After completion of chemotherapy and assessment of response, all patients should undergo surgery. Surgery should be performed 1-14 days after completion (i.e. day 21) of the last chemotherapy cycle. If the tumor is still too large for breast conservation, modified radical mastectomy is recommended. The patient can be offered autologous or heterologous reconstructive surgery. Sentinel node biopsy is allowed to be the only dissected axillary lymph node in patients with a pathological complete response and non involved sentinel node. Surgical reports will be collected and analyzed centrally.

The excised breast tissue should be examined by the pathologist according to guidelines given in the appendix. Histology reports will be collected and analyzed centrally.

Radiotherapy should be applied according to guidelines. Further postoperative systemic treatment is not planned except tamoxifen 20 mg p.o. daily for 5 years (starting after surgery) to patients with positive estrogen and/or progesterone receptors unless there is a contraindication for the use of tamoxifen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained and documented according to the local regulatory requirements prior to beginning specific protocol procedures.
* Complete baseline documentation sent to SKM CRS.
* Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration is not sufficient. Incisional biopsy is not allowed. In case of bilateral cancer the investigator has to decide prospectively which side will be evaluated for the primary endpoint.
* Tumor lesion in the breast with a palpable size of > 2 cm in maximum diameter. The leasion has to be measurable in two-dimensions by sonography. In case of inflammatory disease the extent of inflammation can be used as measurable lesion. The following tumor stages are eligible:

  * Palpable breast tumor size of > 2 cm without involvement of the skin or muscle or evidence of inflammatory disease (T2-3). Clinical N0-2. (Study population I)
  * Primary tumor with clinical involvement of skin or muscle or clinically evidence of inflammatory breast cancer (T4 a-d) or clinical N3 including supraclavicular nodes. (Study population II). In patients with multifocal or multicentric breast cancer, the largest lesion should be measured.
* Age > 18 years.
* Karnofsky Performance status index > 80%.
* Normal cardiac function must be confirmed by LVEF or shortening fraction (echocardiography or MUGA scan respectively) within 3 months prior to registration. The result must be above the normal limit of the institution.
* Laboratory requirements (within 14 days prior to registration):

  * Hematology:

    * Neutrophils > 2.0 x 109/L and
    * Platelets > 100 x 109/L and
    * Hemoglobin > 10 g/dL
  * Hepatic function:

    * Total bilirubin < 1 x UNL and
    * ASAT (SGOT) and ALAT (SGPT) < 2.5 x UNL and
    * Alkaline phosphatase < 5 UNL. Patients with ASAT and/or ALAT > 1.5 x UNL associated with alkaline phosphatase > 2.5 x UNL are not eligible for the study.
  * Renal function:

    * Creatinine < 175 µmol/L (2 mg/dL)
* Tissue block centrally available for further biological tests.
* Negative pregnancy test (urine or serum) within 14 days prior to registration for all women of childbearing potential.
* Complete staging work-up within 3 months prior to registration. All patients must have bilateral mammography, breast ultrasound, breast MRI (optional), chest X-ray (PA and lateral), abdominal ultrasound and/or CT scan, and bone scan. In case of positive bone scan, bone X-ray is mandatory. Other tests may be performed as clinically indicated.
* Patients must be available and compliant for treatment and follow-up. Patients registered on this trial must be treated and followed up at the participating center which can be the Principal or the Co- Investigator's site.

Exclusion Criteria:

* Early breast cancer with a tumor size of < 2 cm measured by palpation.
* Patients with low or moderate risk. These patients are defined as having none of the following risk factors: Age < 36 years, cT> 5cm, ER and PR negative, cN+, or Grade III.
* Evidence of distant metastasis.
* Prior chemotherapy for any malignancy.
* Pregnant or lactating patients. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures during study treatment.
* Pre-existing motor or sensory neuropathy of a severity > grade 2 by NCI criteria.
* Other serious illness or medical condition:

  * previous malignant disease with a disease-free survival of less than 5 years (except CIS of the Cervix and non-melanomatous skin cancer.
  * congestive heart failure or unstable angina pectoris, previous history of myocardial infarction within 1 year prior to study entry, uncontrolled arterial hypertension or high-risk uncontrolled arrhythmias.
  * history of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent.
  * active uncontrolled infection.
  * active peptic ulcer, unstable diabetes mellitus.
* Chronic treatment with corticosteroids unless initiated > 6 months prior to study entry and at low dose (</= 20 mg methylprednisolone or equivalent).
* Concurrent treatment with sex hormones. Prior treatment must be stopped before study entry.
* Definite contraindications for the use of corticosteroids.
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.
* Concurrent treatment with any other anti-cancer therapy.
* Known hypersensitivity reaction to one of the investigational compounds or incorporated substances.
* Male patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2014 (Actual)
Dates: Start 2002-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Determination of pCR rates | 2010
  To determine the iRR rate of 4 cycles of docetaxel, doxorubicin and cyclophosphamide (TAC) and of 4 cycles of vinorelbine and capecitabine (NX) (TAC-NX) as a salvage treatment

SECONDARY OUTCOMES:
To determine the toxicity and compliance to each arm | 2010
  Any grade III/IV toxicity (NCI-CTC Version 2.0) Premature treatment discontinuation
To determine the breast conservation rate in each arm | 2010
  Any breast conservation without reconstruction
To determine the disease-free and overall survival in each arm | 2010
  Any disease related event (recurrence, metastasis) and/or death after primary diagnosis
To determine the specificity and sensitivity of a presurgical core biopsy to predict the degree of pathologic tumor regression | 2010
  No microscopic evidence of residual viable tumor cells (invasive or non-invasive) in all resected specimens of the breast

CONTACTS AND LOCATIONS:
Overall Officials: Gunter von Minckwitz, MD, Principal Investigator — GBG Forschungs GmbH

REFERENCES:
- [Result] von Minckwitz G, Kummel S, Vogel P, Hanusch C, Eidtmann H, Hilfrich J, Gerber B, Huober J, Costa SD, Jackisch C, Loibl S, Mehta K, Kaufmann M; German Breast Group. Neoadjuvant vinorelbine-capecitabine versus docetaxel-doxorubicin-cyclophosphamide in early nonresponsive breast cancer: phase III randomized GeparTrio trial. J Natl Cancer Inst. 2008 Apr 16;100(8):542-51. doi: 10.1093/jnci/djn085. Epub 2008 Apr 8. PMID 18398097
- [Result] Costa SD, Loibl S, Kaufmann M, Zahm DM, Hilfrich J, Huober J, Eidtmann H, du Bois A, Blohmer JU, Ataseven B, Weiss E, Tesch H, Gerber B, Baumann KH, Thomssen C, Breitbach GP, Ibishi S, Jackisch C, Mehta K, von Minckwitz G. Neoadjuvant chemotherapy shows similar response in patients with inflammatory or locally advanced breast cancer when compared with operable breast cancer: a secondary analysis of the GeparTrio trial data. J Clin Oncol. 2010 Jan 1;28(1):83-91. doi: 10.1200/JCO.2009.23.5101. Epub 2009 Nov 9. PMID 19901111
- [Result] Rody A, Karn T, Gatje R, Ahr A, Solbach C, Kourtis K, Munnes M, Loibl S, Kissler S, Ruckhaberle E, Holtrich U, von Minckwitz G, Kaufmann M. Gene expression profiling of breast cancer patients treated with docetaxel, doxorubicin, and cyclophosphamide within the GEPARTRIO trial: HER-2, but not topoisomerase II alpha and microtubule-associated protein tau, is highly predictive of tumor response. Breast. 2007 Feb;16(1):86-93. doi: 10.1016/j.breast.2006.06.008. Epub 2006 Sep 28. PMID 17010609
- [Derived] Leichsenring J, Vladimirova V, Solbach C, Karn T, Ataseven B, Sinn BV, Barinoff J, Muller V, Blohmer JU, Schem C, Engels K, Marme F, Fisseler-Eckhoff A, Fasching PA, Stickeler E, van Mackelenbergh M, Denkert C, Stenzinger A, Loibl S, Groschel S. EVI1 expression in early-stage breast cancer patients treated with neoadjuvant chemotherapy. BMC Cancer. 2022 Oct 5;22(1):1040. doi: 10.1186/s12885-022-10109-1. PMID 36195836
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Lindner JL, Loibl S, Denkert C, Ataseven B, Fasching PA, Pfitzner BM, Gerber B, Gade S, Darb-Esfahani S, Sinn BV, Huober J, Engels K, Tesch H, Karn T, Pommerenke F, Liedtke C, Untch M, Muller V, Rack B, Schem C, von Minckwitz G. Expression of secreted protein acidic and rich in cysteine (SPARC) in breast cancer and response to neoadjuvant chemotherapy. Ann Oncol. 2015 Jan;26(1):95-100. doi: 10.1093/annonc/mdu487. Epub 2014 Oct 29. PMID 25355716
- [Derived] Darb-Esfahani S, von Minckwitz G, Denkert C, Ataseven B, Hogel B, Mehta K, Kaltenecker G, Rudiger T, Pfitzner B, Kittel K, Fiedler B, Baumann K, Moll R, Dietel M, Eidtmann H, Thomssen C, Loibl S. Gross cystic disease fluid protein 15 (GCDFP-15) expression in breast cancer subtypes. BMC Cancer. 2014 Jul 28;14:546. doi: 10.1186/1471-2407-14-546. PMID 25070172
- [Derived] von Minckwitz G, Blohmer JU, Costa SD, Denkert C, Eidtmann H, Eiermann W, Gerber B, Hanusch C, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Kummel S, Paepke S, Schneeweiss A, Untch M, Zahm DM, Mehta K, Loibl S. Response-guided neoadjuvant chemotherapy for breast cancer. J Clin Oncol. 2013 Oct 10;31(29):3623-30. doi: 10.1200/JCO.2012.45.0940. Epub 2013 Sep 3. PMID 24002511
- [Derived] Sinn BV, von Minckwitz G, Denkert C, Eidtmann H, Darb-Esfahani S, Tesch H, Kronenwett R, Hoffmann G, Belau A, Thommsen C, Holzhausen HJ, Grasshoff ST, Baumann K, Mehta K, Dietel M, Loibl S. Evaluation of Mucin-1 protein and mRNA expression as prognostic and predictive markers after neoadjuvant chemotherapy for breast cancer. Ann Oncol. 2013 Sep;24(9):2316-24. doi: 10.1093/annonc/mdt162. Epub 2013 May 9. PMID 23661292
- [Derived] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812